CLINICAL TRIAL: NCT02093949
Title: Substrate Ablation Guided by Automatic High Density Mapping for the Treatment of Atrial Fibrillation
Brief Title: Substrate Ablation Guided by High Density Mapping in Atrial Fibrillation
Acronym: SUBSTRATE-HD
Status: Completed | Type: Observational
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Principal Investigator, SEITZ JULIEN, MD , Cardiologist Rythmologist, Hospital St. Joseph, Marseille, France
Other Study IDs: SUBSTRATE-HD
Record Dates: First submitted 2014-03-14; First posted 2014-03-21 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Studied: Between September 2013 and July 2014, 105 patients were enrolled in 3 centers performing routinely Atrial Fibrillation ablation guided by spatio-temporal electrogram dispersion without pulmonary vein Isolation
  Interventions: Procedure: Routine substrate ablation without pulmonary vein Isolation
- Control: The validation set included a cohort of 47 patients with symptomatic drug-refractory AF who underwent ablation using a conventional approach.
  Interventions: Procedure: Routine conventional ablation with pulmonary vein Isolation

INTERVENTIONS:
Procedure: Routine substrate ablation without pulmonary vein Isolation
  Groups: Studied
Procedure: Routine conventional ablation with pulmonary vein Isolation
  Groups: Control

SUMMARY:
To evaluate a new AF Substrate mapping method based on automatic high density CFAE detection with a multipolar catheter (Pentaray) and the " SCI 30-40 " setting of CARTO CFAE algorithm.

DETAILED DESCRIPTION:
This study is observational :

This substrate ablation method is performed routinely in the centers involved in the study so, patients were not assigned by the investigators to undergo a specific procedure because of the study, in all cases patient would have beneficiate from this substrate mapping ablation method.

We assessed procedural and follow up outcomes of this subatrate ablation group and compared them with an historical control group undergoing conventional ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patient from 18 to 85, with AF* (paroxysmal, and persistent AF) and indication of AF ablation (including redos)* *In accordance with the recommendation of European Society of Cardiology (2010).

Exclusion Criteria:

* organized atrial activity (Atrial tachycardia or Flutter)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient from 18 to 85, with AF* (paroxysmal, and persistent AF) and indication of AF ablation (including redos)*
  *In accordance with the recommendation of European Society of Cardiology (2010).
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julien Seitz, MD, Principal Investigator — St Joseph hospital Marseille
Locations (3):
- France (3):
  - Hopital Saint Joseph, Marseille
  - CHU, Nice
  - Institut Mutualiste de Montsouris, Paris

REFERENCES:
- [Derived] Seitz J, Bars C, Theodore G, Beurtheret S, Lellouche N, Bremondy M, Ferracci A, Faure J, Penaranda G, Yamazaki M, Avula UM, Curel L, Siame S, Berenfeld O, Pisapia A, Kalifa J. AF Ablation Guided by Spatiotemporal Electrogram Dispersion Without Pulmonary Vein Isolation: A Wholly Patient-Tailored Approach. J Am Coll Cardiol. 2017 Jan 24;69(3):303-321. doi: 10.1016/j.jacc.2016.10.065. PMID 28104073

RESULTS

PARTICIPANT FLOW:
Groups:
- Substrate Ablation: Between September 2013 and July 2014, 105 patients with AF were prospectively enrolled at three centers performing substrate ablation (without pulmonary vein isolation) routinely
- Historical Control: The validation set included a cohort of 47 patients with symptomatic drug-refractory AF who underwent ablation using a conventional approach
Period: Overall Study
Arm/Group | Substrate Ablation | Historical Control
Started | 105 | 47
Completed | 105 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Substrate Ablation: Study population (n=105) Between September 2013 and July 2014, 105 patients were enrolled in 3 centers performing routinely Atrial Fibrillation ablation guided by spatio-temporal electrogram dispersion without pulmonary vein Isolation.
- Historical Control: Validation set (n=47) The validation set included a cohort of 47 patients with symptomatic drug-refractory AF who underwent ablation using a conventional approach
- Total: Total of all reporting groups
Arm/Group | Substrate Ablation | Historical Control | Total
Number analyzed (Participants) | 105 | 47 | 152
Age, Continuous [Mean (Standard Deviation); unit: year] | 63 (11) | 58 (11) | 61 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 12 | 37
  Male | 80 | 35 | 115
Paroxysmal AF [Number; unit: participants] | 24 | 9 | 33
Nonparoxysmal AF [Number; unit: participants] | 81 | 38 | 119
Structural heart disease [Number; unit: participants] | 38 | 14 | 52
Hypertension [Number; unit: participants] | 48 | 20 | 68
Diabetes [Number; unit: participants] | 13 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patient With Atrial Fibrillation Termination at the End of the Procedure
Description: percentage of patient in sinus rhythm or in atrial tachycardia at the end of the procedure
Time Frame: up to 240 min
Measure: Number; unit: Percentage of participants
Groups:
- Substrate Ablation: Between September 2013 and July 2014, 105 patients were enrolled in 3 centers performing routinely Atrial Fibrillation ablation guided by spatio-temporal electrogram dispersion without pulmonary vein Isolation
Arm/Group | Substrate Ablation | Historical Control
Number analyzed (Participants) | 105 | 47
Percentage of participants | 95 | 60

2. Secondary Outcome: % of Patients With Sinus Rhythm Conversion During the Procedure
Time Frame: 180 min
Measure: Number; unit: % of participants
Arm/Group | Substrate Ablation | Historical Control
Number analyzed (Participants) | 105 | 47
% of participants | 71 | 26

3. Secondary Outcome: Radiofrequency Time (Min)
Time Frame: up to 300 min
Measure: Number; unit: min
Arm/Group | Substrate Ablation | Historical Control
Number analyzed (Participants) | 105 | 47
min | 49.1 | 84.6

4. Secondary Outcome: Percentage of Patients Free From Atrial Fibrillation 18 Months Post Ablation
Description: % of patients in sinus rhythm or in atrial tachycardia assessed by ECG and/ot 24h-Holter monitoring and clinical examination during follow-up.
Time Frame: 18 Months post ablation
Population: Group Substrate ablation long term follow-up n= 96/105: 9 patients (8.6%) did not complete the follow up; 1 patient died (myocardial infarction) and 8 were lost because of relocation.
  Historical control long term follow-up group n=44/47: 3 patients dropped out during the blanking period (1 died of heart failure and 2 relocated)
Measure: Number; unit: % of participants
Groups:
- Substrate Ablation Long Term Follow Up: Out of the 105 patients included in the substrate ablation arm, only 96 were included in the long term follow-up group.
  9 patients (8.6%) did not complete the follow up: 1 patient died 2 months before the end of follow-up (myocardial infarction) and 8 were lost to follow-up because of relocation.
- Historical Control Long Term Follow-up: Out of the 47 patients included in the validation set arm, only 42 finished the 18-mlonth follow-up. 2 patients were lost to follow-up
  Population at the end of follow up : 3 patients dropped out during the blanking period (1 died of heart failure and 2 relocated)
Arm/Group | Substrate Ablation Long Term Follow Up | Historical Control Long Term Follow-up
Number analyzed (Participants) | 96 | 44
% of participants | 89 | 42

5. Secondary Outcome: Number of Patients With Major Adverse Events During and up to 18 Months After Procedure
Description: Adverse events
Time Frame: 18 months post ablation
Population: as for outcome 4
Measure: Number; unit: participants
Groups:
- Substrate Ablation Long Term Follow-up: Out of the 105 patients included in the substrate ablation arm, only 96 were included in the long term follow-up group.
  9 patients (8.6%) did not complete the follow up: 1 patient died 2 months before the end of follow-up (myocardial infarction) and 8 were lost to follow-up because of relocation.
- Historical Control Long Term Follow-up: Population at the end of follow up : 3 patients dropped out during the blanking period (1 died of heart failure and 2 relocated)
Arm/Group | Substrate Ablation Long Term Follow-up | Historical Control Long Term Follow-up
Number analyzed (Participants) | 96 | 44
participants | 1 | 1

6. Secondary Outcome: Maximum Sustained AF Duration
Description: duration of the longest AF epiodes in months before ablation
Time Frame: from first AF episode to baseline
Measure: Number; unit: months
Arm/Group | Substrate Ablation | Historical Control
Number analyzed (Participants) | 105 | 47
months | 12.2 | 19.4

7. Secondary Outcome: Mean LA Volume
Description: Left Atrial volume before ablation in ml
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Substrate Ablation
Number analyzed (Participants) | 105
ml | 168 (45)

8. Secondary Outcome: Spontaneous AF at the Beginning of the Procedure
Description: Spontaneous AF at the beginning of the procedure
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Substrate Ablation
Number analyzed (Participants) | 105
Participants | 65

ADVERSE EVENTS:
Time Frame: from ablation to 18 month follow up
Groups:
- Substrate Ablation: Study population (n=105)
- Historical Control: Validation set (n=47)
Arm/Group | Substrate Ablation | Historical Control
Serious Adverse Events (participants affected / at risk) | 1/105 | 0/47
Other Adverse Events (participants affected / at risk) | 0/105 | 0/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Substrate Ablation (N=105) | Historical Control (N=47)
Redo Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) — occuring few months after initial ablation during second ablation procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No